CLINICAL TRIAL: NCT04127084
Title: Effects of SGLT2 Inhibition Treatment on Different Levels of Albuminuria in Patients With Type 2 Diabetes: a Prospective Interventional Study
Brief Title: Effects of SGLT2 Inhibition Treatment on Different Levels of Albuminuria in Patients With Type 2 Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongshan Hospital Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20191005
Record Dates: First submitted 2019-10-08; First posted 2019-10-15 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Type 2 Diabetes; Diabetic Nephropathy
Keywords: Type 2 diabetes; Diabetic Nephropathy; Albuminuria; SGLT2 inhibitor
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Nephropathies; Albuminuria

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- normal albuminuria (Experimental): baseline urinary albumin creatinine ratio [UACR]< 30 mg/g
  Interventions: Drug: SGLT2 Inhibition
- moderately increased albuminuria (Experimental): baseline UACR 30~300 mg/g
  Interventions: Drug: SGLT2 Inhibition
- severely increased albuminuria (Experimental): baseline UACR>300mg/g
  Interventions: Drug: SGLT2 Inhibition
- blank Comparator (No Intervention): normal participant

INTERVENTIONS:
Drug: SGLT2 Inhibition — Dapagliflozine 5-10 mg once daily tablet treatment or Empagliflozin10 mg once daily tablet treatment or Canagliflozin 100 mg once daily tablet treatment
  Other Names: Dapagliflozine,Empagliflozin,Canagliflozin
  Arms: moderately increased albuminuria; normal albuminuria; severely increased albuminuria

SUMMARY:
Diabetic kidney disease has become the leading cause for ESRD worldwide.Albuminuria is a major risk factor for progression of diabetic nephropathy. SGLT2 inhibitors are the first antiglycaemic drugs with direct renoprotection, which are thought to protect the kidneys by lowering albuminuria, stimulating urinary glucose excretion ,reducing systemic blood pressure, while simultaneously improving multiple other risk factors in a glucose-independent manner. However, the precise mechanisms behind the renal beneficial effect of SGLT2 inhibitors are not entirely elucidated, although ongoing outcome trials will confirm these findings. This study is to assess the impact of three months of treatment with SGLT2 Inhibitions on different levels of albuminuria in patients with type 2 diabetes and to evaluate the effects of SGLT2 inhibition treatment on markers for podocyte damage , renal fibrosis, inflammation，oxidative stress and renin-angiotensin- aldosterone system.

DETAILED DESCRIPTION:
Objective: The primary objective is to assess the impact of three months of treatment with SGLT2 Inhibition on Different levels of Albuminuria in Patients With type 2 diabetes and to seek the relationship of this influences to relevant risk markers in the pathology of diabetic renal disease.

Design: prospective ，intervention， case-controlled , single center study. Treatment period: 12 weeks. Patient population: 60 patients with type 2 diabetes recruited from Zhongshan Hospital Xiamen University in accordance with the study in- and exclusion criteria.

Intervention: Dapagliflozine 10 mg once daily tablet treatment or Empagliflozin10 mg once daily tablet treatment or Canagliflozin 100 mg once daily tablet treatment. Endpoints: Primary outcome: evaluate the effects of SGLT2 inhibition treatment on on urinary albuminuria, kidney function and eGFR .

Secondary endpoints To assess the effect of SGLT2 inhibition on markers for podocyte damage , renal fibrosis, inflammation，oxidative stress and renin-angiotensin- aldosterone system。 Timeframe: Recruiting planned from October 2019, inclusion over the following 12 months. Last patient is expected to be completed October 2020. Data analysis completed December 2020, publication autumn 2021.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients between 18 -80 years of age with a diagnosis of type 2 diabetes (WHO criteria).
2. HbA1c of 7-11 %
3. eGFR equal to or above 45 ml/min/1.73 m2
4. The Trial included 20 normal albuminuria (Urinary albumin creatinine ratio [UACR]< 30 mg/g, with 20 moderately increased albuminuria UACR 30~300 mg/g, and 20 severely increased albuminuria UACR>30 0mg/g (in ≥2 out 3 morning spot urine collections prior to enrolment ).at baseline.
5. Patients who agree to receive treatment with SGLT2 inhibitors.
6. Patients must be on current stable hemodynamic profile , without dehydration.
7. Patients must be on current stable antiglycaemic treatment with oral drugs (OAD) or insulin 4 weeks before start of study drug and throughout study duration.
8. Patients must be on stable antihypertensive treatment (not include renin-angiotensin system blocking treatment) 4 weeks before start of study drug and throughout study duration.

Exclusion Criteria:

1. type 1 diabetes
2. Patients who suffer from recent acute complications including diabetic ketoacidosis and hyperglycaemic hyperosmolar coma, which may be at risk for dehydration.
3. Patients with hypertension who are not on stable antihypertensive treatment
4. urinary tract or reproductive tract acute infection
5. impaired liver function, defined as aspartate aminotransferase (AST) >3x upper limit of normal (ULN) and/or alanine aminotransferase (ALT) >3x ULN
6. History of unstable or rapidly progressing renal disease
7. impaired renal function ,eGFR: <45 mL/min (calculated by MDRD formula)
8. Ongoing cancer treatment
9. Recent Cardiovascular Events in a patient:

   9.1. Acute Coronary Syndrome (ACS) within 2 months prior to enrolment 9.2.Hospitalization for unstable angina or acute myocardial infarction within 2 months prior to enrolment9. 3. Acute Stroke or TIA within two months prior to enrolment 9. 4. Less than two months post coronary artery revascularization
10. Congestive heart failure defined as New York Heart Association (NYHA) class IV, unstable or acute congestive heart failure..
11. Pregnant or breastfeeding patients
12. smoker.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Change in urinary albuminuria | Up to 12 weeks
  a clean-catch 24- hour urine sample and spot urine sample were collected to assess urinary albuminuria,which will be evaluated at week 0, and at end study week 12 (+/- 1 week)
Change in eGFR | Up to 12 weeks
  eGFR was calculated by modified glomerular filtration rate estimating equation for Chinese patients with chronic kidney disease.
change in nephrin | Up to 12 weeks
  To assess effect of SGLT2 inhibition intervention on glomerular podocyte injury by detecting the expression of renal nephrin.
change in TGF-β1 | Up to 12 weeks
  To assess effect of SGLT2 inhibition intervention on glomerular and tubulointerstitial fibrosis by detecting the expression of TGF-β1
change in IL-6 | Up to 12 weeks
  To assess effect of SGLT2 inhibition intervention on inflammation biomarkers by detecting the levels of interleukin-6.
change in TNFα | Up to 12 weeks
  To evaluate the effects of SGLT2 inhibition treatment on inflammation, biomarkers by detecting the levels of tumor necrosis factor alpha.
changes of AGEs | Up to 12 weeks
  To evaluate the effects of SGLT2 inhibition treatment on oxidative stress index, the changes of AGEs.
changes of 8-OH-dG | Up to 12 weeks
  To evaluate the effects of SGLT2 inhibition treatment on oxidative stress index by detecting the levels of 8-OH-dG.
  Urinary 8-OH-dG concentrations were assayed using a competitive enzyme-linked immunosorbent assay

SECONDARY OUTCOMES:
Change in uric acid | Up to 12 weeks
  To evaluate the levels of serum uric acid before and after SGLT2 inhibition treatment.
Change in aldosterone | Up to 12 weeks
  To evaluate the levels of aldosterone before and after SGLT2 inhibition treatment.
Change in rennin | Up to 12 weeks
  To evaluate the levels of rennin before and after SGLT2 inhibition treatment
Change in angiotensin | Up to 12 weeks
  To evaluate the levels of angiotensin before and after SGLT2 inhibition treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yi-lin Zhao, principal, Study Director — Zhongshan Hospital Xiamen University
Locations (1):
- Zhongshan Hospital Xiamen University, Xiamen, Fujian, China

REFERENCES:
- [Derived] Zeng XC, Tian Y, Liang XM, Wu XB, Yao CM, Chen XM. SGLT2i relieve proteinuria in diabetic nephropathy patients potentially by inhibiting renal oxidative stress rather than through AGEs pathway. Diabetol Metab Syndr. 2024 Feb 16;16(1):46. doi: 10.1186/s13098-024-01280-5. PMID 38365853
- [Derived] Tian Y, Chen XM, Liang XM, Wu XB, Yao CM. SGLT2 inhibitors attenuate nephrin loss and enhance TGF-beta1 secretion in type 2 diabetes patients with albuminuria: a randomized clinical trial. Sci Rep. 2022 Sep 20;12(1):15695. doi: 10.1038/s41598-022-19988-7. PMID 36127497